CLINICAL TRIAL: NCT05162573
Title: Tolerability of Concurrent EBRT + Lu-PSMA for Node-positive Prostate Cancer (PROQURE-1)
Brief Title: EBRT + Lu-PSMA for N1M0 Prostate Cancer
Acronym: PROQURE-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: UMC Utrecht (Other); Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M21PQ1; 2020-005577-27 (EudraCT Number); NL75976.031.21 (Other: Centrale Commissie Mensgebonden Onderzoek (CCMO))
Record Dates: First submitted 2021-10-07; First posted 2021-12-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Prostatic Neoplasm
Keywords: Lu-PSMA; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto

STUDY DESIGN:
Intervention Model Description: Multicenter prospective phase I study investigating standard of care treatment for node-positive prostate cancer (7 weeks EBRT and 3 years ADT) complemented with 1 or 2 concurrent cycles of systemic 177Lu-PSMA-617 delivered in week 2 (and 4) of EBRT. The tolerability of adding 177Lu-PSMA-617 will be evaluated using a Bayesian Optimal Interval (BOIN) dose-escalation design based on the occurrence of grade 3 acute toxicity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EBRT + 3 GBq Lu-PSMA (Experimental)
  Interventions: Drug: 177Lu-PSMA-617; Radiation: EBRT
- EBRT + 6 GBq Lu-PSMA (Experimental)
  Interventions: Drug: 177Lu-PSMA-617; Radiation: EBRT
- EBRT + 9 GBq Lu-PSMA (Experimental)
  Interventions: Drug: 177Lu-PSMA-617; Radiation: EBRT
- EBRT + 2x7.4 GBq Lu-PSMA (Experimental)
  Interventions: Drug: 177Lu-PSMA-617; Radiation: EBRT

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — Dose-escalation of 177Lu-PSMA-617 (3, 6, 9 or 2x7.4 GBq) combined with external beam radiotherapy (EBRT)
Radiation: EBRT — External Beam Radiotherapy

SUMMARY:
The PROQURE project aims to provide prostate cancer patients with more cure and better quality of life. The first part of this project (PROQURE-1) aims to explore an innovative combined modality treatment strategy for patients with node-positive prostate cancer (N1M0). The current standard of care for these patients, external beam radiotherapy (EBRT) of the prostate and regional pelvic nodes combined with 2-3 years androgen deprivation therapy (ADT), leads to suboptimal tumor control while inducing significant and potentially persistent toxicity. To overcome this, the current locoregional treatment is complemented with systemic Lutetium-177-PSMA radioligand therapy in a phase I study, with the aim to achieve better tumor control while potentially reducing or obviating ADT and its associated toxicity for future patients.

DETAILED DESCRIPTION:
Rationale: In the past, prostate cancer patients with nodal metastases (clinically N1M0) were not considered for curative treatment, based on the hypothesis that these patients are affected by systemic disease. Today, patients with primary diagnosed N1M0 prostate cancer increasingly receive curative intent high-dose external beam radiotherapy (EBRT) to the prostate and regional nodes combined with up to 3 years androgen deprivation therapy (ADT). This aggressive and lengthy multimodal treatment can achieve long-term disease-free and overall survival, but it also comes with significant toxicity and failure rates of up to 47% within 5 years with locoregional recurrence within radiotherapy fields and/or distant progression. A new strategy is needed to (1) enhance EBRT to better control macroscopic tumor in the prostate and involved nodes, (2) better treat undetected microscopic disease inside and outside EBRT fields, and (3) potentially reduce or obviate the long use of ADT with its toxicity and associated poor quality of life. Radioligand therapy (RLT) with Lutetium-177 labeled PSMA-ligands (177Lu-PSMA-617) can selectively deliver radiation dose to both macroscopic and microscopic tumor locations throughout the body, with limited systemic toxicity. Based on radiobiologic considerations, the hypothesis is that complementing EBRT with concurrent 177Lu-PSMA-617 can provide synergistic anti-tumor effects, without prolonging overall treatment time and with limited toxicity. The feasibility of this innovative use of "RLT as the ultimate radiosensitizer for EBRT" now needs to be explored.

Objective: Primary: To determine the maximum tolerated dose (MTD) of 1 or 2 cycles 177Lu-PSMA-617 when given concurrent with EBRT+ADT. Secondary: To demonstrate acceptable late toxicity at 6 months, superior dosimetric efficacy, anti-tumor efficacy at 6 months, feasibility of QoL evaluation and favorable pharmacokinetics.

Study design: Multicenter prospective phase I dose-escalation study, using a BOIN design, with 4 dose levels for 177Lu-PSMA-617 and a maximum of 24 patients.

Study population: Patients with primary diagnosed prostate cancer, clinical stage T2-T4N1M0 based on MRI and PSMA PET/CT, with a PSMA-positive index tumor within the prostate and involved nodes all within EBRT fields (highest node below the level of the aortic bifurcation).

Intervention: Standard of care treatment (EBRT of prostate and pelvic nodes with concurrent ADT) is complemented with 1 or 2 concurrent cycles dose-escalated 177Lu-PSMA-617 in week 2 (and 4).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participation in the study involves one day hospitalization per administration with IV catheter and administration of 3, 6 or 9 or 2x7.4 GBq 177Lu-PSMA-617 in week 2 (and week 4) of EBRT, and during the week after each administration 3 SPECT/CT scans from pelvis to head for dosimetry and 11 blood samples for pharmacokinetics. Patient receives additional radiation exposure from 177Lu-PSMA-617, which comes with a low risk for acute toxicity (infusion reaction, nausea, vomiting), low risk for late toxicity (temporary salivary gland function loss), a maximum of one of two days hospitalization in isolation, and after discharge about 2 weeks radiation safety measures at home. These disadvantages are considered acceptable for patients with node-positive prostate cancer, in the scope of potential improvements in tumor control with associated benefits in survival and QoL, for included patients as well as for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer;
* cT2-4, partly determined by MRI;
* N1, determined by LND/SNP and/or PSMA PET/CT;
* iM0, determined by PSMA PET/CT;
* Accepted for curative intent treatment with EBRT of the prostate and regional nodes + 3y ADT;
* Visually PSMA-positive primary tumor and nodes, largest lesion ≥ average liver uptake;
* WHO performance score 0-1;
* Age > 18 years;
* For patients who have partners of childbearing potential: Willingness to use a method of birth control with adequate barrier protection during the study and for 6 months after the study drug administration; and
* Signed written informed consen

Exclusion Criteria:

* Inability to comply to study procedures;
* Inability to adhere to radiation safety measures in hospital or at home;
* Inability to undergo the required biodistribution scans;
* Prior or current malignant disease with potential impact on treatment outcome or survival;
* Prior treatment with EBRT;
* Prior treatment with ADT, already initiated >1 month before the start of EBRT;
* Prior treatment with radionuclide therapies, 177Lu-PSMA-617 or other;
* Reduced bone marrow reserve (Hb<6 mmol/L, Leukocytes<2.5 10E9/L, or Platelets<100 10E9/L not older than 1 month before start of EBRT);
* Reduced renal function (GFR < 60 not older than 1 month before start of EBRT);
* Reduced salivary gland function (history of prior salivary gland disease); or
* Miction problems requiring pre-treatment with ADT.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | from start of EBRT until 3 months after EBRT
  The maximum tolerated dose (MTD) of the 4 selected doses of Lu-PSMA (3, 6, 9 and 2x7.4 GBq) when administered in combination with EBRT.

SECONDARY OUTCOMES:
Dose-limiting-toxicity (DLT) | From start of EBRT until 3 months after EBRT
  grade 3 toxicity according to CTCAE v5.0
Late toxicity | 6 months after EBRT
  grade 3 toxicity according to CTCAE v5.0
Anti-tumor efficacy | 6 months after EBRT
  PSA response

CONTACTS AND LOCATIONS:
Overall Officials: Wouter V Vogel, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (2):
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] van der Sar ECA, Braat AJAT, van der Voort-van Zyp JRN, van der Veen BS, van Leeuwen PJ, de Vries-Huizing DMV, Hendrikx JMA, Lam MGEH, Vogel WV. Tolerability of concurrent external beam radiotherapy and [177Lu]Lu-PSMA-617 for node-positive prostate cancer in treatment naive patients, phase I study (PROQURE-I trial). BMC Cancer. 2023 Mar 23;23(1):268. doi: 10.1186/s12885-023-10725-5. PMID 36959540